CLINICAL TRIAL: NCT01923129
Title: Prospective Study Investigating Optimal Duration of Indwelling Urinary Catheter Following Infraperitoneal Colorectal Surgery and Role of Postoperative Alpha Blockade
Brief Title: Optimal Duration of Indwelling Urinary Catheter Following Pelvic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Fleshner MD, Widjaja Chair in Colorectal Surgery, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00029210
Record Dates: First submitted 2013-07-29; First posted 2013-08-15 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-01

CONDITIONS: Urinary Retention
Keywords: indwelling catheter; foley; duration
MeSH Terms: conditions — Urinary Retention | interventions — Population Groups; Prazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 24 hour postop catheter removal (Experimental): group will receive the study medication prazosin ( 1 mg PO) 6 hours prior to catheter discontinuation (24 hours postoperatively)
  Interventions: Drug: Prazosin given 6 hours prior to catheter removal in the 24 hour group
- 72 hour postoperative catheter removal (No Intervention): catheter removed on postoperative day 3 (72 hours postoperatively)

INTERVENTIONS:
Drug: Prazosin given 6 hours prior to catheter removal in the 24 hour group — Prazosin given orally (1 mg) 6 hours prior to catheter removal (hour 18 postoperatively)
  Other Names: Minipress; Vasoflex; Pressin; Hypovase
  Arms: 24 hour postop catheter removal

SUMMARY:
There is no general agreement about the optimal duration of postoperative urinary drainage, with relevant literature reporting durations ranging from 1 to 10 days. The available research supporting the routine use of prolonged catheterization is limited and studies investigating early removal following infraperitoneal colorectal surgery have largely been underpowered to form valid practice conclusions. The aim of the investigators study is to determine whether a postoperative colorectal patient can safely have an indwelling catheter removed on postoperative day one (24 hours following surgery) with the addition of a study medication (prazosin), without a statistically significant difference in the incidence of urinary retention compared to the standard, accepted approach of delayed removal (72 hours postoperatively). Patients undergoing laparoscopic and open pelvic colorectal surgery below the peritoneal reflection for both benign and malignant conditions will be randomized into two groups: group one will have the catheter removed on postoperative day 3 (72 hours postoperatively) Group 2 will have a dose of the alpha-blocker prazosin given 6 hours prior to catheter removal and will have the urinary catheter removed on postoperative day 1 (24 hours postoperatively).

DETAILED DESCRIPTION:
The available research supporting the routine use of prolonged catheterization is limited and studies investigating early removal following infraperitoneal colorectal surgery have largely been underpowered to form valid practice conclusions. In the era of multimodal recovery algorithms emphasizing early diet advancement, ambulation, and shorter hospital length of stay, unnecessarily prolonging catheterization may interfere with many of these objectives. An indwelling urinary catheter interferes with early patient mobilization potentially lengthening hospitalization and subjects patients to an increased risk of urinary tract infection. A study of 2,355 consecutive patients undergoing primary colorectal cancer resection via laparotomy found an overall prevalence of postoperative urinary retention of 5.5%, however, those patients undergoing low pelvic surgery experience an almost 16% incidence in urinary retention.

Postoperative urinary catheter drainage after infraperitoneal colorectal surgery is commonly practiced, assuming some degree of nerve damage to the superior hypogastric plexus at the sacral promontory or of the nervi erigentes at the pelvic side wall resulting from pelvic dissection, causing transient or permanent dysfunction of the lower urinary tract. It has been believed that this intraoperative damage to the pelvic autonomic nerves may be associated with early postoperative acute urinary retention, and justifies an indwelling urinary catheter for several days following infraperitoneal pelvic surgery. However, there is no general agreement about the optimal duration of postoperative urinary drainage, with relevant literature reporting durations ranging from 1 to 10 days.

Prolonged indwelling urinary catheter has been associated with increased risk of urinary tract infections, with the risk of bacteriuria between 3 and 10% per day when catheterized, with the risk of urinary tract infection increasing by 5% to 10% per catheter day after the second day of catheterization. The incidence of urinary tract infections after anorectal surgery and 5 days of catheterization has been shown to range between 42% and 60%. Higher mortality rates have been reported in hospitalized patients who developed urinary tract infection after indwelling catheterization with the incidence of bacteremia after single catheterization reported to be as high as 8%.

The optimal duration of urinary drainage after infraperitoneal colorectal surgery is unknown. Based on the autonomic mechanisms of micturition in relation to the striated muscle fibers of the external urethral sphincter, alpha blockade has been studied as a potential intervention to reduce the incidence of re-catheterization. A large Cochrane Database reviewed their role in five randomized trials, with four trials favoring alpha blockade over placebo. Furthermore, the side-effect profile of alpha-blockade was low and compared favorably to placebo.

Prior studies have suggested urinary bladder catheter drainage removed on postoperative day one following pelvic surgery may be safe and decrease the incidence of urinary tract infection. However, the study was underpowered to detect meaningful conclusions. A larger study investigating the optimal duration of urinary drainage concluded that removing the catheter one day postoperatively in patients undergoing infraperitoneal colorectal surgery is appropriate, unless a low rectal carcinoma is present or lymph node metastatic disease is present. The investigators wish to further substantiate this evidence and introduce the positive findings associated with alpha-blockade in minimizing the need for re-catheterization.

The investigators therefore propose a prospective, controlled randomized trial to compare the effects of 1 day's transurethral catheterization after infraperitoneal surgery with an alpha blockade medication compared to those of 3 days of catheterization, with acute urinary retention as a primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Able to freely give written informed consent to participate in the study and have signed the Informed Consent Form;
2. Males or females, >18 years of age inclusive at the time of study screening;
3. American Society of Anesthesiologists (ASA) Class I-III;
4. Infraperitoneal colorectal surgery (open and/or laparoscopic);
5. Elective Surgery

Exclusion Criteria:

1. Mentally incompetent or unable or unwilling to provide informed consent or comply with study procedures;
2. Children <18;
3. No perioperative antibiotics;
4. Past or current urinary tract malignancy;
5. Urinary catheter inserted before surgery;
6. Chronic kidney insufficiency with Creatinine> 2
7. Diagnosis of benign prostatic hyperplasia
8. Chronic urinary infections
9. Neurogenic bladder
10. History of enterovesical fistula
11. Pregnancy
12. Prior surgery of the lower urinary tract
13. Epidural
14. Perioperative ureteral stents

After randomization:

1. Catheter pulled out inadvertently;
2. Postoperative complications requiring prolonged monitoring of urine output
3. Postoperative complications requiring early reoperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2012-11-30 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Fleshner, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246
- [Derived] Patel DN, Felder SI, Luu M, Daskivich TJ, N Zaghiyan K, Fleshner P. Early Urinary Catheter Removal Following Pelvic Colorectal Surgery: A Prospective, Randomized, Noninferiority Trial. Dis Colon Rectum. 2018 Oct;61(10):1180-1186. doi: 10.1097/DCR.0000000000001206. PMID 30192326

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 subjects were excluded.
Period: Overall Study
Arm/Group | 24 Hour Postop Catheter Removal | 72 Hour Postoperative Catheter Removal
Started | 71 | 71
Completed | 71 | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 24 Hour Postop Catheter Removal | 72 Hour Postoperative Catheter Removal | Total
Number analyzed (Participants) | 71 | 71 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.07 (16.9) | 45.6 (17.8) | 44.8 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 37 | 68
  Male | 40 | 34 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 58 | 59 | 117
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 71 | 71 | 142
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 24.4 (4.9) | 23.78 (4.2) | 24.1 (9.1)
American Society of Anesthesiologists Physical Status Classification [Count of Participants; unit: Participants] — ASA I A normal healthy patient
  ASA II A patient with mild systemic disease Mild diseases only without substantive functional limitations.
  ASA III A patient with severe systemic disease Substantive functional limitations; One or more moderate to severe diseases.
  ASA IV A patient with severe systemic disease that is a constant threat to life
  Participants
    1 | 3 | 1 | 4
    2 | 51 | 51 | 102
    3 | 15 | 19 | 34
    4 | 2 | 0 | 2
Surgery Indication [Count of Participants; unit: Participants]
  inflammatory bowel disease | 55 | 48 | 103
  Cancer | 11 | 19 | 30
  Prolapse | 3 | 2 | 5
  Other | 2 | 2 | 4
Type of Surgery [Count of Participants; unit: Participants]
  IPAA | 53 | 41 | 94
  LAR | 12 | 14 | 26
  Rectopexy | 3 | 3 | 6
  Other | 3 | 13 | 16
Surgical drain [Count of Participants; unit: Participants]
  Yes | 66 | 57 | 123
  No | 5 | 14 | 19
intraoperative intravenous fluids [Mean (Standard Deviation); unit: milliliters] — This is crystalloids received via intravenous access during surgery
  milliliters | 2855.6 (803) | 2948.6 (857) | 2901 (192)
intraoperative estimated blood loss [Mean (Standard Deviation); unit: milliliters] — A clinical estimate of surgical blood loss determined by the lead surgeon and anesthesiologist after the conclusion of the case.
  milliliters | 182 (82) | 201 (99) | 192 (91)
OR time [Mean (Standard Deviation); unit: minutes] | 282 (66) | 301 (61) | 292 (191)
peri-operative blood transfusion [Count of Participants; unit: Participants]
  yes | 1 | 5 | 6
  no | 70 | 66 | 136
Total mesorectal excision [Count of Participants; unit: Participants] — Total mesorectal excision (TME) employs a precise, sharp dissection between the visceral and parietal layers of the endopelvic fascia to ensure en bloc removal of the perirectal areolar tissue, including the lateral and circumferential margins of the mesorectal envelope, lymphatics, and vascular/perineural tumor deposits with the primary rectal cancer. TME also preserves the autonomic nerves and reduces the risk of presacral bleeding.
  Participants
    yes | 18 | 16 | 34
    no | 53 | 55 | 108
neoadjuvant chemotherapy [Count of Participants; unit: Participants]
  yes | 5 | 6 | 11
  no | 66 | 65 | 131
intravenous pain medications on post-operative day one [Mean (Standard Deviation); unit: milligrams of hydromorphone] — in the immediate 24 hours following surgery, the total amount of intravenous narcotics consumed by the patient was recorded and collected. All intravenous narcotics were converted into equivalent milligrams of hydromorphone.
  milligrams of hydromorphone | 4.6 (1.73) | 4.8 (1.65) | 4.7 (1.7)
mean pain score [Mean (Standard Deviation); unit: units on a scale] — This is a 1-10 scale Pain 0: No pain at all, you feel perfectly normal. Pain 1: Very light barely noticeable pain Pain 2: Minor pain, Discomforting Pain 3: Tolerable pain Pain 4: Distressing, Strong, deep pain Pain 5: Very Distressing, Strong, deep, piercing pain Pain 6: Intense Pain deep, piercing pain so strong it seems to partially dominate your senses Pain 7: Very Intense Pain Pain 8: Horrible Pain: so intense you can no longer think clearly at all Pain 9: Excruciating, so intense you cannot tolerate Pain 10: Unimaginable Pain, so intense you will go unconscious shortly.
  units on a scale | 3.84 (1.09) | 3.91 (1.09) | 3.87 (1.1)
The tumor, node, metastasis (TNM) staging system of the combined American Joint Committee on Cancer [Count of Participants; unit: Participants] — This is a staging system from stage 0 (best, no tumor) to stage 4 (worst, metastatic disease).
  T = tumor stage (T1 is best and invades submucosa, T2 invades muscularis, T3 invades pericolorectal tissues, T4 is worst and adherent to other organs N = nodal stage (N0 negative nodes is best, N+ positive nodes is worse) M = metastases stage (M0 no metastases is best, M+ metastases is worse)
  The categories are:
  0: T0, N0, M0
  1. T1-T2, N0, M0
  2. T3-T4, N0, M0
  3. Any T stage, N+, M0
  4. Any T or N stage, M+
  Participants
    0 | 57 | 51 | 108
    1 | 8 | 10 | 18
    2A | 4 | 3 | 7
    2B | 0 | 0 | 0
    2c | 0 | 1 | 1
    3a | 1 | 3 | 4
    3b | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Urinary Retention
Description: Acute urinary retention will be defined as catheter discontinuation with inability to void 6 hours post-removal, or void with post-void residual greater than 200 cc of urine.
Time Frame: Postoperative day 1 or postpoperative 3 depending on group randomization
Measure: Count of Participants; unit: Participants
Arm/Group | 24 Hour Postop Catheter Removal | 72 Hour Postoperative Catheter Removal
Number analyzed (Participants) | 71 | 71
Participants | 6 | 7

2. Secondary Outcome: Number of Participants With a Symptomatic Urinary Tract Infection
Description: Urinary tract infection defined as symptomatic urinary complaints such as dysuria, with urinalysis consistent with infection.
Time Frame: During 1 week of hospitalization (prior to discharge)
Measure: Count of Participants; unit: Participants
Arm/Group | 24 Hour Postop Catheter Removal | 72 Hour Postoperative Catheter Removal
Number analyzed (Participants) | 71 | 71
Participants | 0 | 8
Statistical Analysis 1: Comparison: 24 Hour Postop Catheter Removal vs 72 Hour Postoperative Catheter Removal; Test type: Non-Inferiority — The primary outcome of interest was the rate of AUR, defined as the number of patients with AUR within each study group. A 15% non-inferiority margin was chosen according to clinical relevance estimation. The expected difference between the two groups was 0%. Non-inferiority analysis was performed by calculation of risk difference and its 95% confidence interval according to Newcombe & Altman; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 72 hours
Description: Methods did not differ from definitions provided by clinicaltrials.gov
Arm/Group | 24 Hour Postop Catheter Removal | 72 Hour Postoperative Catheter Removal
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/71
Other Adverse Events (participants affected / at risk) | 6/71 | 0/71
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24 Hour Postop Catheter Removal (N=71) | 72 Hour Postoperative Catheter Removal (N=71)
Dizziness (Cardiac disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-11-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT01923129/Prot_000.pdf
  • Statistical Analysis Plan (2012-11-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT01923129/SAP_001.pdf